CLINICAL TRIAL: NCT07371442
Title: Effectiveness of Audiovisual Distraction and Acuapoint Stimulation on Anxiety and Pain Perception During Tooth Extraction in Children: A Randomized Controlled Clinical Study.
Brief Title: Effect of AV Distraction and Acuapoint Stimulation in Pediatric Extraction on Pain and Anxiety
Acronym: AV Acupoint
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A03012024PP
Record Dates: First submitted 2026-01-11; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Tooth Extraction; Local Anesthesia; Anxiety; Pain
Keywords: Audiovisual; acuapoint; acupressure; TSD; pain; anxiety; tooth extraction
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dental story (Experimental): A dental video story will be presented to patient using an iPad device connected to a noise cancellation headphone.
  Interventions: Device: Audiovisual
- Aculief (Experimental): Aculief acupressure device will be placed on the LI4 Point which is located on the hand between the thumb and index finger, also described as the depression where the index finger and thumb bone go apart. The LI4 point will be identified in each patient by asking the patient to adduct the thumb and index finger. The duration will be 5 minutes before LA administration. to patients
  Interventions: Device: Acualief
- TSD (Experimental): This group will be treated using Tell-show-do technique
  Interventions: Behavioral: TELL SHOW DO

INTERVENTIONS:
Device: Acualief — Aculief acupressure device will be placed on the LI4 Point (figure 1) which is located on the hand between the thumb and index finger, also described as the depression where the index finger and thumb bone go apart. The LI4 point will be identified in each patient by asking the patient to adduct the thumb and index finger. The duration will be 5 minutes before LA administration.
  The administration of local anesthesia in all groups will be achieved by 1.8 ml of 2% Lidocaine with 1/100,000 epinephrine using a 30-gauge long needle
  Arms: Aculief
Device: Audiovisual — A dental video story will be presented to the patient using an iPad device connected to a noise cancellation headphone.
  Arms: dental story
Behavioral: TELL SHOW DO — This group will be treated using Tell-show-do technique
  Arms: TSD

SUMMARY:
The aim of this study is to evaluate the effectiveness of audiovisual distraction and acuapoint stimulation on anxiety and pain perception during tooth extraction in children.

ELIGIBILITY:
Inclusion Criteria:

* 1- Children with behavior rating score 2,3 according to Frankl's behavior rating scale.

  2- Children aged 5-8 years requiring primary tooth extraction. 3- Healthy children free of systemic diseases

Exclusion Criteria:

* 1- Children with special health care needs.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 69 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Will be measured 5 minutes before LA , immediately before extraction and immediately after extraction The total VPT score was obtained by summing the values across all eight panels, with higher scores indicating greater levels of anxiety (range: 0-8).
  Anxiety will be measured by A) Pulse oximeter: Pulse oximeter was used to observe the physiological functions like heart rate and SpO₂.
  B) Venham's picture test: the child was presented with eight different cards. Each card held two pictures-a representation of the child expressing anxiety along with another representation of the same child in a relaxed mood. The child was asked to point out the picture in each pair that resembled how he/she was feeling. There was also an order in which the pictures had to be presented. Assigning the image depicting anxiety the score of 1 and the relaxed image the score of 0 helped in the coding process.

SECONDARY OUTCOMES:
Pain of the patient | Will be evaluated immediately after the local anesthesia and tooth extraction using Wong Baker FACES Pain rating scale, ranging from a no pain (score 0) to one showing severe pain (score 5)
  will be evaluated by Wong baker FACES pain scale which is consist of six faces numbered ordinary from 0 to 5. ranging from a no pain (score 0) to one showing severe pain (score 5)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Mansoura university, Al Mansurah, Egypt